CLINICAL TRIAL: NCT03771417
Title: Resistance Exercise and Low-Intensity Physical Activity Breaks in Sedentary Time to Improve Skeletal Muscle and Cardiometabolic Health in Older Adults-REALPA Breaks in Sedentary Time Pilot Study
Brief Title: Resistance Exercise and Low-Intensity Physical Activity Breaks in Sedentary Time to Improve Muscle and Cardiometabolic Health
Acronym: REALPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University and A&M College (Other)
Collaborators: Pennington Biomedical Research Center (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Brian Irving, Associate Professor, Louisiana State University and A&M College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-026; R21AG058181 (NIH)
Record Dates: First submitted 2018-12-07; First posted 2018-12-11 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Aging; Sarcopenia; Disability Physical; Cardiovascular Diseases; Insulin Resistance; Diabetes Mellitus
MeSH Terms: conditions — Sarcopenia; Cardiovascular Diseases; Insulin Resistance; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resistance Exercise (Experimental): Exercise Intervention: Participants will be asked to complete supervised resistance exercise 2 days per week.
  Interventions: Behavioral: Exercise Intervention
- RE plus Low Intensity Physical Activity (Experimental): Exercise Intervention: Participants will be asked to complete supervised resistance exercise 2 days per week and regular unsupervised low intensity physical activity breaks in sedentary time 5 days per week [6x10 min breaks/d at 2 metabolic equivalents (METS) or ~30-40% peak oxygen consumption (VO2 peak), ~500 kcal/wk above resting metabolism].
  Interventions: Behavioral: Exercise Intervention
- RE plus Moderate IntensityExercise (Active Comparator): Exercise Intervention: Participants will be asked to complete supervised RE 2 days per week and supervised calorically matched moderate intensity physical activity 3 days per week (50 min/session at 4 METS (~60-75% VO2 peak), ~500 kcal/week above resting metabolism).
  Interventions: Behavioral: Exercise Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — The use of exercise to improve muscle and cardiometabolic health in older adults.

SUMMARY:
What are the effects of resistance exercise (RE) alone or RE plus low intensity physical activity (LPA) breaks in sedentary time (ST) on skeletal muscle health in older adults?

What are the effects of resistance exercise (RE) alone or RE plus low intensity physical activity (LPA) breaks in sedentary time (ST) on skeletal cardiometabolic health in older adults?

DETAILED DESCRIPTION:
Although awareness of the detrimental impact that sedentary behavior has on skeletal muscle and cardiometabolic health has increased over the last 20 years, more than 60% of older adults remain sedentary for greater than 8 hours per day. Moreover, 80% to 90% of adults 60 years of age or older do not meet the current public health guidelines for aerobic exercise (AE) or resistance exercise (RE) based physical activity (PA). Collectively, these adverse health behaviors contribute to the development of multiple chronic medical conditions commonly afflicting older adults, including type 2 diabetes, cardiovascular disease, sarco/dynapenia, frailty, and premature mortality. Emerging evidence suggests that breaking up sedentary time with light intensity PA (LPA) improves muscle and cardiometabolic health. Recent data also suggest that RE combined with moderate intensity AE effectively improves muscle and cardiometabolic health in older adults. However, the impact that RE combined with LPA breaks in sedentary time has on muscle and cardiometabolic health in older adults remains unknown. The overall objective of this pilot study is to determine the effect of 16 weeks of RE alone or RE combined with LPA breaks in sedentary time on muscle and cardiometabolic health.

ELIGIBILITY:
Inclusion Criteria:

1. Are capable and willing to give written informed consent, and understand exclusion criteria
2. 65-80 years of age inclusive
3. Body Mass Index (BMI) between 18.5-34.9 kg/m2, inclusive
4. Physically inactive determined by self-report
5. Stable medical therapy for allowable medications for 30 days defined as:

   1. No addition or removal of a medication
   2. No change in dosage of a medication
6. Having no life-threatening conditions or diseases
7. Willing to allow researchers to use data, bio-specimens (blood and muscle tissue), and images (e.g., magnetic resonance imaging) for research purposes after study participation is completed
8. At least 2 weeks post-completion of the COVID19 vaccine regimen. a. Acceptable proof of vaccine includes a completed vaccine card and/or letter from a healthcare provider indicating the date that the COVID19 vaccine was completed.

Exclusion Criteria:

1. Nursing home resident
2. Physically Active:

   a. > 100 min/wk of moderate OR > 50 min/wk vigorous intensity PA
3. Saint Louis University Mental State (SLUMS) score < 21
4. Evidence or self-report history of deep vein thrombosis, pulmonary embolism, cardiovascular, peripheral vascular, cerebral vascular, pulmonary, or renal disease
5. Evidence or self-report history of type 1 or 2 diabetes mellitus
6. Evidence or self-report history of a bleeding disorder
7. Evidence or self-report history of recurrent vasovagal episodes
8. Evidence or self-report history of severe depression, Schizophrenia, bipolar disease
9. Evidence or self-report history of mobility disability requiring a walker, wheel chair, or inability to walk across a small room.
10. Evidence or self-report history of orthopedic limitations that would preclude them from participation in a dynamic exercise program
11. Evidence or self-report history of severe arthritis (either osteoarthritis or rheumatoid arthritis) that would preclude them from participation in a dynamic exercise program
12. Evidence or self-report of history untreated thyroid dysfunction.
13. Weight loss of > 10% in the last 3 months prior to screening
14. History of weight loss surgery.
15. Use of medications known to influence study outcomes, such as:

    1. Insulin
    2. Oral antidiabetic medications (e.g., metformin)
    3. Corticosteroids
    4. Beta-blockers

    c. Anticoagulants
16. Allergy to lidocaine
17. Active smoking
18. Current consumption of > 14 alcoholic drinks per week based on self-report
19. Regular participation in resistance or aerobic exercise training within 3 months of initial screening
20. Absolute Contraindication to Exercise as Defined by the American College of Sports Medicine,16 including:

    1. Resting diastolic blood pressure > 100 mm Hg
    2. Resting systolic blood pressure > 180 mm Hg
    3. Resting heart rate > 100 beats per min
21. Having a body weight greater than 440 pounds
22. Having medical implants such as a pacemaker or metal joint replacements
23. Having tattoos or permanent makeup completed <30 days prior to the visit
24. Recent (past 3 months) cancer diagnosis, undergoing immunotherapy, taking immune suppressants
25. Presence of allergies or infections requiring antibiotics within the past 14 days
26. Recent (past 3 months) major surgery on the abdomen, pelvis, or lower extremities
27. Any other condition that in the judgement of the Principal Investigator and/or the Medical Director of this protocol may interfere with study participation and adherence to the protocol.
28. Evidence or self-report history of severe depression in the last 5 years.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Irving, PhD, Principal Investigator — Louisiana State University and A&M College
Locations (2):
- United States (2):
  - Lousiana State University, Baton Rouge, Louisiana
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana

REFERENCES:
- [Derived] Marazzato F, McCarthy C, Field RH, Nguyen H, Nguyen T, Shepherd JA, Tinsley GM, Heymsfield SB. Advances in digital anthropometric body composition assessment: neural network algorithm prediction of appendicular lean mass. Eur J Clin Nutr. 2024 May;78(5):452-454. doi: 10.1038/s41430-023-01396-3. Epub 2023 Dec 23. PMID 38142263
- [Derived] McCarthy C, Tinsley GM, Yang S, Irving BA, Wong MC, Bennett JP, Shepherd JA, Heymsfield SB. Smartphone prediction of skeletal muscle mass: model development and validation in adults. Am J Clin Nutr. 2023 Apr;117(4):794-801. doi: 10.1016/j.ajcnut.2023.02.003. Epub 2023 Feb 8. PMID 36822238
- [Derived] Wong MC, Bennett JP, Leong LT, Tian IY, Liu YE, Kelly NN, McCarthy C, Wong JMW, Ebbeling CB, Ludwig DS, Irving BA, Scott MC, Stampley J, Davis B, Johannsen N, Matthews R, Vincellette C, Garber AK, Maskarinec G, Weiss E, Rood J, Varanoske AN, Pasiakos SM, Heymsfield SB, Shepherd JA. Monitoring body composition change for intervention studies with advancing 3D optical imaging technology in comparison to dual-energy X-ray absorptiometry. Am J Clin Nutr. 2023 Apr;117(4):802-813. doi: 10.1016/j.ajcnut.2023.02.006. Epub 2023 Feb 14. PMID 36796647

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 24 participants were enrolled in the present study, 23 participants were randomized. 1 participant did not complete baseline testing.
Groups:
- RE Plus Moderate Intensity Exercise: Exercise Intervention: Participants will be asked to complete supervised RE 2 days per week and supervised calorically matched moderate intensity physical activity 3 days per week (50 min/session at 4 METS (~60-75% VO2 peak), ~500 kcal/week above resting metabolism).
  Exercise Intervention: The use of exercise to improve muscle and cardiometabolic health in older adults.
Period: Overall Study
Arm/Group | Resistance Exercise | RE Plus Low Intensity Physical Activity | RE Plus Moderate Intensity Exercise
Started | 7 | 8 | 8
Completed | 6 | 7 | 8
Not Completed | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Covid-19 Shutdown | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: One participant in the resistance training group withdrew from the study due to time conflict, and one participant in the RE plus Low Intensity Physical Activity was lost to follow-up due to shutdown of campus during the beginning of the covid 19 pandemic.
Groups:
- Total: Total of all reporting groups
Arm/Group | Resistance Exercise | RE Plus Low Intensity Physical Activity | RE Plus Moderate IntensityExercise | Total
Number analyzed (Participants) | 7 | 8 | 8 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (2.9) | 70.4 (3.9) | 69.5 (5.0) | 70.0 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 5 | 16
  Male | 2 | 2 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 4
  White | 5 | 7 | 7 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Skeletal Muscle Strength
Description: The investigators will determine the change from baseline in skeletal muscle strength. These measurements will be performed at baseline and following 16 weeks of exercise training using isokinetic dynamometry and 1 repetition maximum testing.
Time Frame: Measured at week 0 (baseline) and week 16
Population: Change is Leg Press 1-RM
Measure: Mean (Standard Error); unit: Change in Lbs
Arm/Group | Resistance Exercise | RE Plus Moderate Intensity Exercise | RE Plus Low Intensity Physical Activity
Number analyzed (Participants) | 6 | 8 | 7
Change in Lbs | 93.9 (17.9) | 50.0 (15.2) | 78.6 (15.2)

2. Primary Outcome: Skeletal Muscle Mass
Description: The investigators will determine the change from baseline in skeletal muscle mass. These measurements will be performed at baseline and following 16 weeks of exercise training using Dual X-Ray Absorptiometry.
Time Frame: Measured at week 0 (baseline) and week 16
Population: Change Appendicular Lean Mass (kg/m^2)
Measure: Mean (Standard Error); unit: Change Appendicular Lean Mass (kg/m^2)
Arm/Group | Resistance Exercise | RE Plus Moderate Intensity Exercise | RE Plus Low Intensity Physical Activity
Number analyzed (Participants) | 6 | 8 | 7
Change Appendicular Lean Mass (kg/m^2) | 0.22 (0.11) | 0.17 (0.10) | 0.27 (0.10)

3. Secondary Outcome: Mitochondrial Function
Description: The investigators will determine the change from baseline in mitochondrial function. These measurements will be performed at baseline and following 16 weeks of exercise training.
Time Frame: Measured at week 0 (baseline) and week 16
Population: Change skeletal muscle oxidative capacity measured using high-resolution respirometry in permeabilized muscle fibers for complex I and II substrates (pyruvate, malate, glutamate, and succinate) expressed as pmols/sec/mg wet weight.
Measure: Least Squares Mean (Standard Error); unit: pmols/sec/mg wet weight
Arm/Group | Resistance Exercise | RE Plus Low Intensity Physical Activity | RE Plus Moderate IntensityExercise
Number analyzed (Participants) | 6 | 7 | 3
pmols/sec/mg wet weight | 27.2 (5.9) | 17.0 (5.4) | 5.9 (8.3)

ADVERSE EVENTS:
Time Frame: During study period, up to 16 weeks
Arm/Group | Resistance Exercise | RE Plus Moderate Intensity Exercise | RE Plus Low Intensity Physical Activity
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resistance Exercise (N=7) | RE Plus Moderate Intensity Exercise (N=8) | RE Plus Low Intensity Physical Activity (N=8)
Fall (Investigations) | 0 (0) | 0 (0) | 1 (1) — One participant fell during a study visit.
Vasovagal (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — One participant experienced a vasovagal syncope episode during one of their strength assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT03771417/Prot_SAP_000.pdf